CLINICAL TRIAL: NCT05146310
Title: Prospective, Multicenter, Non-comparative Clinical Investigation to Support Safety & Effectiveness of I.SPACE® Ophthalmic Viscosurgical Device
Brief Title: Prospective, Multicenter, Non-comparative Clinical Investigation to Support Safety & Effectiveness of I.SPACE®
Acronym: PROMIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Collaborators: International Clinical Trials Association (Other); Inferential (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A01486-35
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Cataract
Keywords: anterior segment of the eye; hyaluronic acid; corneal endothelium; surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: One group of patient treated with I.SPACE® (instilled in the anterior chamber of the eye and adjusted according to the volume of the aqueous humour)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated eye (Experimental): Eye is treated at Baseline visit (V1)
  Interventions: Device: I.SPACE®

INTERVENTIONS:
Device: I.SPACE® — I.SPACE® is a viscoelastic sodium hyaluronate gel use as a surgical aid in ophthalmic anterior segment surgery by maintaining the intraocular space and protecting the corneal endothelium.
  The baseline injection is performed at V1. The volume of product to use will be at the Investigator discretion, and will be completely removed after surgery.

SUMMARY:
I.SPACE® is a hyaluronic acid injectable gel CE (European Conformity) marketed since 2010. It is indicated for use as a surgical aid in ophthalmic anterior segment surgery. The aim is to protect the corneal endothelium and maintains the intraocular space.The product should be instilled in the anterior chamber of the eye and adjusted according to the volume of the aqueous humour.

In this study, 80 patients aged from 18 to 84 years' old at inclusion, who have at least one eye with cataract (mild to moderate severity) based on subjective ophthalmic examination by the investigator, who have given his/her informed consent and meet all the eligibility criteria, will be enrolled.

Subjects will come to a total of 7 visits over a period of 3 months. Protection of corneal endothelium (Mean percent change of CEC density) after baseline injection will be assessed. Surgeon's satisfaction during cataract surgery, mean change in Intraocular Pressure (IOP), percentage of eyes with IOP spikes ≥ 30mm mmHg, corneal thickness, intraocular inflammation, Mean Snellen monocular Uncorrected Distance Visual Acuities (UCDVA), Best Corrected Distance Visual Acuities (BCDVA) and safety will be also assessed.

DETAILED DESCRIPTION:
PROMIR is a prospective, multicenter, non-comparative post-marketing study of a class IIb medical device (medical device regulatory classification IIb).

This uncontrolled open-label study investigates the efficacy and safety of I.SPACE® in corneal endothelium protection and intraocular space maintain.

The study duration is 3 months with a screening visit (V0) up to 14 days before injection, the baseline visit (injection of I.SPACE®), V1) and 5 follow-up visits after 6 hours, 24 hours, 7 days, 30 days and 90 days (V1' to V5). It is envisaged to enroll 80 patients with planned cataract surgery for at least 1 eye in France to obtain at least 68 evaluable patients, which will be monitored over 3 months after baseline injection of I.SPACE® .

The primary endpoint is defined as the mean percent change of CEC density at 3 months (90 days) post-operation (V5) from Baseline (V0). The effectiveness of I.SPACE® will be demonstrated if the CEC density loss is statistically non-superior to a pre-specified threshold of 10% (non-inferiority to -10%).

Surgeon's satisfaction after cataract surgery (questionnaire) will be evaluated at V1.

Protection of corneal endothelium (Mean percent change of CEC density) will be also assessed at V4.

Mean change in Intraocular Pressure (IOP), percentage of eyes with IOP spikes ≥ 30mm mmHg, intraocular inflammation and safety will be assessed at all timepoints.

Corneal thickness will be assessed at V2,V3 and V5. Mean Snellen monocular Uncorrected Distance Visual Acuities (UCDVA), Best Corrected Distance Visual Acuities (BCDVA) and ocular symptoms will be assessed at V2, V3, V4 and V5.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged from 18 to 84 years' old at inclusion.
* Having at least one eye with cataract (mild or moderate severity) based on subjective ophthalmic examination by the investigator.
* Informed of the clinical investigation and having given freely and expressly his/her informed consent.
* Affiliated to a health social security system.
* Female of childbearing potential should use a medically accepted contraceptive regimen since at least 12 weeks before screening visit.

Exclusion Criteria:

In terms of population

* Pregnant or breastfeeding women or planning a pregnancy during the clinical investigation.
* Participating at the same time in another clinical investigation or is in an exclusion period of one.
* Deprived of their freedom by administrative or legal decision or under guardianship.
* Known hypersensitivity to one of the investigational medical device (IMD) ingredients.
* One-eyed patients.

In terms of associated pathology

* Pre-existing :

  * Glaucoma,
  * severe myopia,
  * diabetic retinopathy,
  * retinal vascular disease,
  * Acute ocular disease or external infection or internal infection or uveitis prior to surgery,
  * Known ocular disease/pathology that may affect visual acuity or that may be expected to require retinal laser treatment or other surgical intervention (other than cataract surgery) during the course of the study.
  * Any causes of compromised aqueous humor outflow.
* History of :

  * Intraocular surgery,
  * ocular trauma,
  * lens pseudoexfoliation capsular syndrome,
  * ocular hypertension > 21 mmHg without treatment
  * chronic or recurrent inflammatory eye disease or a congenital ocular anomaly such as Marfan's Syndrome
* Endothelial cell density at baseline less than 2000 cells/mm2 or poor quality photograph of preoperative endothelial cells (all reasons including corneal abnormalities).
* Any abnormalities that prevented reliable Goldmann applanation tonometry.
* Eyes with Axial Length (AL) >25 mm or < 20 mm or eyes with small pupil diameter, pathologic miosis or pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils);

Relating to previous and ongoing treatments:

* Patient currently treated with Tamsulosine and other alpha 1 antagonist or psychotics

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Mean percent change of Corneal Endothelium Cells (CEC) density | 3 months (90 days)
  Mean percent change of CEC density at 3 months (90 days) post-operation from Baseline. The effectiveness of I.SPACE® will be demonstrated if the CEC density loss is statistically non-superior to a pre-specified threshold of 10% (non-inferiority to -10%).

SECONDARY OUTCOMES:
Intraocular space maintenance evaluation | Baseline (surgery)
  Evaluation of the intraocular space maintenance (questionnaire) using a 4-point scale, assessed by the surgeon, at Baseline. The 4-point scale contains the following categories : "Not at all", "Slightly"; "Very much" and "Extremely".
Surgeon's satisfaction evaluation | Baseline (surgery)
  Evaluation of surgeon's satisfaction after cataract surgery (questionnaire) using a 4-point scale assessed by the surgeon, at Baseline. Each cataract surgery stage should be evaluated with a 4-point scale containing the following categories : "Full chamber maintained ", "Work space maintained"; "Shallow" and "flat".
Mean percent change of CEC density | 30 days
  Mean percent change of CEC density evaluated from baseline to 30 days.
Mean change in Intraocular Pressure (IOP) | 6 hours, 24 hours, 7 days, 30 days and 90 days.
  Mean change in IOP, measured by Goldmann applanation tonometry, from baseline to 6 hours, 24 hours, 7 days, 30 days and 90 days.
Percentage of eyes with IOP spikes ≥ 30 millimeter of mercury (mmHg) | 6 hours, 24 hours, 7 days, 30 days and 90 days.
  Percentage of eyes with IOP spikes ≥ 30mmHg, measured by Goldmann applanation tonometry, at 6 hours, 24 hours, 7 days, 30 days, and 90 days.
Corneal thickness evaluation | 24 hours, 7 days and 90 days.
  Corneal thickness, evaluated at 24 hours, 7 days and 90 days.
Intraocular inflammation evaluation | 6 hours, 24 hours, 7 days, 30 days and 90 days.
  Intraocular inflammation, evaluated by slit-lamp examination at 6 hours, 24 hours, 7 days, 30 days and 90 days.
Mean Snellen monocular Uncorrected Distance Visual Acuities (UCDVA), Best Corrected Distance Visual Acuities (BCDVA) and ocular symptoms | 24 hours, 7 days, 30 days and 90 days.
  UCDVA and BCDVA under photopic lighting conditions and ocular symptoms, at 24 hours, 7 days, 30 days and 90 days. Ocular symptoms will be subjectively assessed by interrogating the patient. If a subject reports a symptoms, the level of severity should be reported.
Report of adverse effects | 90 days
  Evaluation of product safety by adverse event collection throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: SANTIAGO Pierre-Yves, Dr, Principal Investigator — Institut Ophtalmologique de l'Ouest Jules Verne
Locations (3):
- France (3):
  - Clinique Ophtalmologique Thiers, Bordeaux
  - Centre rétine Gallien, Bordeaux
  - Vision Sud, Marseille